CLINICAL TRIAL: NCT02265120
Title: Primary Care Providers' Views and Understanding of Current Recommended Guidelines for Cervical Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Lavona Lewis, Teaching Professor of Public Policy and Director of Undergraduate Programs, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-14-00447
Record Dates: First submitted 2014-09-30; First posted 2014-10-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- primary care providers by region (Experimental): A questionnaire will be given to a randomized sample of primary care providers who care for patients in the 194 federally designated regions of Primary Care provider shortage within California will be studied.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — The Questionnaire aims to evaluate based on the responses if providers don't uniformly agree with the new guidelines, if they can't interpret them correctly, and or if they have personal biases towards the older guidelines based upon prior training, personal experience, financial incentives, etc.

SUMMARY:
Significant developments have led to a dramatic change in recommendations for cervical cancer screening. The understanding that the Human Papilloma Virus (HPV) is the cause of nearly 100% of cervical cancer cases and the development of new technologies for detection of HPV DNA at time of cervical cancer screening, has produced changes in preventive healthcare policy for this condition. In an unprecedented event, the American College of Obstetrics and Gynecology, the American Cancer Society and the U.S. Preventive Services Task Force recommended dramatic and unified changes in screening utilizing this new framework. No studies of significance have evaluated (since guideline change in 2013), whether primary care providers find the new recommendations authoritative and believe in them, or whether providers understand implementation of these new guidelines given the many decades of contradictory and differing recommendations. For this study, the opinions of primary care providers who care for patients in the 194 federally designated regions of Primary Care provider shortage within California will be studied. Using the California Medical Board database of licensed providers, a questionnaire will be mailed to a random subset. It is anticipated that the analysis will show varying contempt, confusion and compliance with new guidelines exists. Understanding these factors will have beneficial health policy implications in terms of overcoming barriers to these cost-effective, less intrusive, and more accurate health policy guidelines in the prevention and early detection of cervical cancer.

DETAILED DESCRIPTION:
Cervical cancer remains a common cause of death and disability among women both within the United States and world-wide. Potential exists for significant prevention and early detection if cervical cancer screening is performed at the correct frequencies, with correct methods, on the appropriate women. Since the development of the Papanicolaou smear (Pap smear), cervical cancer screening has been recommended as a component of preventative healthcare for women. The tradition of an annual pap smear remains a common component of American medicine. For over four decades, controversy has existed as to the optimal method and timing of cervical cancer screening. The result has been great confusion amongst providers.

Significant developments have led to a dramatic change in recommendations for cervical cancer screening. The understanding that the Human Papilloma Virus (HPV) is the cause of nearly 100% of cervical cancer cases and the development of new technologies for detection of HPV DNA at time of cervical cancer screening, has produced changes in preventive healthcare policy for this condition. In an unprecedented event, the American College of Obstetrics and Gynecology, the American Cancer Society and the U.S. Preventive Services Task Force recommended dramatic and unified changes in screening utilizing this new technology: In healthy women, A: do not start screening prior to age 21, B: screen every 3 years between ages 21-29, C: screen only every 5 years between ages 30-65, and D: stop any further screening for cervical cancer after 65. This significant reduction in the number of cervical cancer screenings is the result of these new technologies for the detection of the HPV virus, as well as evidence-based findings on the lack of risk for cancer in women who test negative for HPV. From a public health policy standpoint, the new recommendations are revolutionary. Whereas a women previously might have received 62 "Pap Smears" between the ages of 18-79, with new recommendations, only 6 cervical cancer screenings would be required over her lifetime.

Understanding these new recommendations and complying with these new unified recommendations would have a dramatic effect on health policy. The current multi-billion dollar cost of annual cervical cancer screening would be dramatically reduced. The time and physical inconvenience of this examination would be lessened. At a time when there is a great shortage of primary care providers (MD's, PA's and NP's) in many parts of the U.S., these dramatically reduced needs for cervical cancer screening might allow primary care providers greater time for more important health policy. No studies of significance have evaluated (since guideline change in 2013), whether primary care providers find the new recommendations authoritative and believe in them, or whether providers understand implementation of these new guidelines given the many decades of contradictory and differing recommendations.

The implications for health policy are significant:

1. To the extent that primary care providers don't believe in the new guidelines, then providers should be educated on the evidence-based rationale from which they were constructed. In other words: to overcome whatever misgivings providers might harbor as to the new recommendations.
2. To the extent that primary care providers believe in the new guidelines, but can't correctly apply them, then health policy would suggest an educational campaign to indicate correct application.
3. To the extent that primary care providers harbor biases, further research to understand and develop strategies to overcome these biases would be indicated.

For this study, the opinions of primary care providers who care for patients in the 194 federally designated regions of Primary Care provider shortage within California will be studied. Using the California Medical Board database of licensed providers, a questionnaire will be mailed to a random subset. The sample will be randomized to include providers in both urban and rural areas of provider shortages, with a spectrum of patients of differing ethnic and economic status. It is anticipated that approximately 5,000 questionnaires will be mailed out with the goal of 1,000 responses.

The study will investigate the following issues: 1) Do primary care providers in these regions believe in these new and dramatically different guidelines? 2) Are the providers able to correctly apply these guidelines in four different clinical vignettes? 3) Do the providers hold a bias which may influence their willingness to follow these new guidelines? It is anticipated that the analysis will show varying contempt, confusion and compliance with new guidelines exists. Understanding these factors will have beneficial health policy implications in terms of overcoming barriers to these cost-effective, less intrusive, and more accurate health policy guidelines in the prevention and early detection of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Primary care providers who care for patients within the 194 federally designated regions of Primary Care provider shortage within California

Exclusion Criteria:

* Outside of federally designated region of Primary Care provider shortage within California

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Primary Health Care Providers Beliefs Regarding Current Cervical Cancer Screening Guidelines | 5 months
  Questionnaire responses to clinical scenarios and assessments of current published clinical guidelines by ACOG, ACS or USPSTF

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Boone, Principal Investigator — University of Southern California
Locations (1):
- USC Sol Price School of Public Policy, Los Angeles, California, United States